CLINICAL TRIAL: NCT06316895
Title: The Clinical Outcomes and Artificial Intelligence Prediction Model of Ultrasound-guided Thermal Ablation for the Treatment of Low-risk Papillary Thyroid Carcinoma
Brief Title: The Clinical Outcomes and Prediction of Thermal Ablation for Low-risk Papillary Thyroid Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Director, Head of Department of Ultrasound, Chinese PLA General Hospital
Other Study IDs: S2023-706
Record Dates: First submitted 2024-02-16; First posted 2024-03-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgery group: patients with low-risk papillary thyroid carcinoma who chose thyroid surgery
  Interventions: Procedure: thyroid surgery
- ablation group: patients with low-risk papillary thyroid carcinoma who chose thermal ablation
  Interventions: Procedure: ultrasound-guided thermal ablation

INTERVENTIONS:
Procedure: thyroid surgery — thyroid lobectomy
  Groups: surgery group
Procedure: ultrasound-guided thermal ablation — radiofrequency ablation; microwave ablation or laser ablation
  Groups: ablation group

SUMMARY:
1. To evaluate the clinical outcomes of ultrasound-guided thermal ablation and thyroid surgery for the treatment of papillary thyroid carcinoma;
2. To develop and validate a artificial intelligence model to predict the outcomes of ultrasound-guided thermal ablation in the treatment of papillary thyroid carcinoma;

ELIGIBILITY:
Inclusion Criteria:

1. patients age between 18 and 80 year old, both sex
2. papillary thyroid carcinoma confirmed by core-needle biopsy or fine-needle aspiration
3. the largest diameter ≤2.0 cm
4. no clinical or imaging evidences of extrathyroidal extension, lymph node metastasis and distant metastasis on ultrasound, nech and chest CT
5. follow-up period ≥12 months,

Exclusion Criteria:

1. patients with convincing evidence of aggressive papillary thyroid carcinoma or other type of thyroid cancer by biopsy
2. history of neck radiation
3. history of thyroid surgery
4. coagulation disorder
5. serious heart, respiratory, liver, or renal failure
6. dysfunction of the vocal cord on the opposite side

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with low-risk papillary thyroid carcinoma who choose surgery or thermal ablation
Sampling Method: Probability Sample
Enrollment: 3772 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of disease progression | more than 5 year
  cervical lymph node metastases, recurrent tumors and persistent tumors

SECONDARY OUTCOMES:
Rate of complications | 1week
  surgery or ablation complications
Rate of tumor disappearance | 2 year
  complete disappearance of ablated tumor on ultrasound and contrast-enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No